CLINICAL TRIAL: NCT02774889
Title: Once 'Stepping On' Ends: Continuing a Group Falls Prevention Program Via the Internet
Brief Title: KOSO (Keep On Stepping On)/ Stepping Online
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-0125; A534255 (Other: UW, Madison); SMPH/MEDICINE/GER-AD DEV (Other: UW, Madison)
Record Dates: First submitted 2016-05-11; First posted 2016-05-17 (Estimated); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Fall Related Injury; Social Isolation
Keywords: Falls Prevention; Stepping On; Health Promotion; Implementation; Health Maintenance
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepping Online (Active Comparator): Stepping On graduates receive Stepping Online, a password-protected continuation website to maintain fall prevention behaviors.
  1. Fall prevention tips
  2. Fall prevention exercise videos noting technique and safety
  3. Guest expert videos and communication with expert
  4. Tools to set exercise goals, reminders and track progress
  5. Fall prevention specialist for feedback and group activities
  6. Discussion and messaging (1:1, small and large group)
  7. Fall prevention resources.
  Interventions: Behavioral: Stepping Online
- Stepping On Usual Care Control (No Intervention): Subjects control workshops in the condition will not have access to Stepping Online.

INTERVENTIONS:
Behavioral: Stepping Online — Stepping Online is a password-protected website with Stepping On graduates, whose groups are randomized to Stepping Online and will have access to and training in a password-protected website. The website includes:
  1. Fall prevention tips
  2. Fall prevention exercise videos with narrations for proper technique and safety precautions
  3. Guest expert videos with online access to the guest expert to ask questions
  4. Tools to set exercise goals, get reminders and track progress
  5. Access to a fall prevention specialist for personal feedback and suggested group homework
  6. Group discussion and messaging (one-to-one and with their fellow Stepping On workshop participants group, or with all Stepping Online participants and leaders)
  7. Fall prevention resources
  Other Names: Keep On Stepping On (KOSO)
  Arms: Stepping Online

SUMMARY:
The overall purpose of this multi-phase study is to develop (Phase 1) and test potential effectiveness and feasibility of Keep On Stepping On (KOSO)/Stepping Online, an online falls prevention maintenance program for Stepping On (SO) graduates in a group randomized trial (Phase 2).

This application refers to effectiveness component of Phase 2, which entails the randomized clinical trial. Phase 1 has been completed. The feasibility component of Phase 2 will entail process evaluation of the Stepping Online intervention group only.

DETAILED DESCRIPTION:
Aim:

This application, for Phase 2 of a larger study, is a 6-month group randomized trial to test the effectiveness of Stepping Online.

Stepping Online (developed in Phase 1) is a continuation website to help Stepping On graduates to:

1. Maintain exercises and fall prevention strategies learned in Stepping On, and
2. Stay connected with other participants and leaders/peer leaders in the 7-week workshop.

Approach:

1. Subject Eligibility:

   1. Stepping On leaders and peer leaders of Milwaukee, Dane, Rock, Adams, Green Lake, Marquette and Waushara Counties during the enrollment window
   2. Stepping On participants/graduates of the above workshops whose leader assesses that they can safely use Stepping Online to exercise at home
2. Recruitment and Consenting:

   1. Leaders/Peer Leaders: County aging unit coordinators will invite leaders to participate in the study and share the names of those who agree with the study research staff. Staff will then explain the study in detail, answer questions, and obtain informed consent from those who agree.
   2. Participants: (1) Research staff will visit participating leader/peer leader workshops to explain the study; (2) leader will distribute a card for participants to agree to a researcher phone call to learn more. They will then share the contact information of those who agree with study research staff; (3) study research staff members will contact and conduct a recruitment interview by phone. They then schedule those who agree to come to the site where the workshop occurred (or another public place that is private and convenient for research subjects) for consenting and baseline measurement.
3. Randomization

   Randomization will occur on the Stepping On workshop level to ensure that leaders, peer leaders and participants are in the same arm. Procedures:
   1. County liaisons, who routinely collect data, will provide participants' education level (without personal identifiers);
   2. Study biostatistician pairs workshops based on above data, as well as geographic location and other data to ensure comparability.
   3. Participants from each designated pair of SO workshops will provide informed consent and participate in baseline measurements
   4. Designated pair of SO workshops will be randomized to the Stepping Online (intervention) or to the usual care Control arm.

   <!-- -->

   1. Intervention arm: Stepping On graduates (and their leaders/peer leaders) will receive the Stepping Online website for 6 months. They can use their own computer or receive a laptop and Internet access (if needed) for the study duration. Research staff will provide 2 in-home training sessions (2 weeks apart) on how to use Stepping Online's fall prevention features (described under the "Arms and Intervention" section). Participants can call the technical support phone line for more help.
   2. Control arm: Stepping On graduates in this arm will not receive Stepping Online.
   3. Neither the intervention nor the control arm subjects will have access to Stepping Online after the 6-month trial.
4. Participants in both study arms will complete measurements at their workshop location or another location that is private and convenient fir subjects at baseline (prior to randomization), and later at 3 and 6 months.

ELIGIBILITY:
List of Inclusion Criteria:

1. Leader/Peer Leader: Leading a SO workshop in Dane, Milwaukee, Rock, Adams, Green Lake, Marquette or Waushara counties during the timeframe prior to the 6-month trial.
2. Stepping On Participants/Graduates: Enrolled in one of the above SO workshops.

In Milwaukee and Dane counties, extra effort will be made to enroll African American Stepping On participants/graduates, who are more likely to have lower income and educational level and to be uninsured than their White counterparts.

List of Exclusion Criteria:

1. Leaders/Peer Leaders:

   1. Not available to participate in Stepping Online for more than 4 weeks out of the 6 months following enrollment
   2. Not in the area at the end of the 6-month trial.
2. Stepping On Participants/Graduates:

   1. Unable participate in Stepping Online for more than 4 weeks out of the 6 months following enrollment
   2. Not assessed to be safe by SO leader to do the online exercise program; not in the area for the 3 month and 6 month evaluations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Mahoney, MD, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clemson L, Fiatarone Singh MA, Bundy A, Cumming RG, Manollaras K, O'Loughlin P, Black D. Integration of balance and strength training into daily life activity to reduce rate of falls in older people (the LiFE study): randomised parallel trial. BMJ. 2012 Aug 7;345:e4547. doi: 10.1136/bmj.e4547. PMID 22872695
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Gustafson DH, Hawkins R, McTavish F, Pingree S, Chen WC, Volrathongchai K, Stengle W, Stewart JA, Serlin RC. Internet-Based Interactive Support for Cancer Patients: Are Integrated Systems Better? J Commun. 2008 Jun;58(2):238-257. doi: 10.1111/j.1460-2466.2008.00383.x. PMID 21804645
- [Background] Clemson L, Cumming RG, Kendig H, Swann M, Heard R, Taylor K. The effectiveness of a community-based program for reducing the incidence of falls in the elderly: a randomized trial. J Am Geriatr Soc. 2004 Sep;52(9):1487-94. doi: 10.1111/j.1532-5415.2004.52411.x. PMID 15341550
- [Background] Mahoney, J. E., Gangnon, R., Clemson, L. M., Gobel, V. L., & Lecey, V. (2012, November). Evaluation of stepping on implementation across Wisconsin. In GERONTOLOGIST (Vol. 52, pp. 479-479). JOURNALS DEPT, 2001 EVANS RD, CARY, NC 27513 USA: OXFORD UNIV PRESS INC.
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the total 157 invitees, 45 enrolled; 112 did not. Of the 112 non-joiners, 53 declined further contact; 16 were not reached; 12 were ineligible, 31 refused.
Groups:
- Stepping Online: Stepping On graduates receive Stepping Online, a password-protected continuation website to maintain fall prevention behaviors.The website includes:
  1. Fall prevention tips
  2. Fall prevention exercise videos with narrations for proper technique and safety precautions
  3. Guest expert videos with online access to the guest expert to ask questions
  4. Tools to set exercise goals, reminders and track progress
  5. Fall prevention specialist for feedback and group activities
  6. Discussion and messaging (1:1, small and large group)
  7. Fall prevention resources.
- Stepping On Usual Care Control: Control Stepping On graduates did not have access to Stepping Online.
Period: Overall Study
Arm/Group | Stepping Online | Stepping On Usual Care Control
Started | 23 | 22
Completed | 21 | 21
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Stepping Online: Stepping On graduates receive Stepping Online, a password-protected continuation website to maintain fall prevention behaviors.
- Stepping On 'Usual Care': Control Stepping On graduates did not have access to Stepping Online.
- Total: Total of all reporting groups
Arm/Group | Stepping Online | Stepping On 'Usual Care' | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (9.04) | 76 (7.35) | 73.6 (8.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 2 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 18 | 21 | 39
  White, Hispanic | 1 | 0 | 1
  African-American | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45
Days Since Last Stepping On Class [Mean (Standard Deviation); unit: days] | 35.9 (6.07) | 37.4 (14.75) | 36.31 (11.37)
Number of Falls in the Past 6 months [Mean (Standard Deviation); unit: falls] | 0.45 (1.12) | 0.50 (0.80) | 0.47 (0.97)
Number of Participants Who Fell At Least 1 in the last 6 months [Count of Participants; unit: Participants] | 6 | 7 | 13
Number of Participants With College Education [Count of Participants; unit: Participants] | 19 | 16 | 35
Number of Married Participants [Count of Participants; unit: Participants] | 14 | 4 | 18
Number of Participants in a City/Suburb [Count of Participants; unit: Participants] | 18 | 13 | 31

OUTCOME MEASURES:

1. Primary Outcome: Change of Number of Falls From Baseline to 6 Months
Description: Number of Falls: monthly calendar self-administered sent and returned via mail
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: falls
Arm/Group | Stepping Online | Stepping On 'Usual Care'
Number analyzed (Participants) | 21 | 21
falls | 0.28 (0.01) | 0.40 (0.00)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On 'Usual Care'; Test type: Superiority; p = 0.55, Fisher Exact; Rate Ratio = 0.72, 95% CI 2-sided [0.27 to 2.57]

2. Secondary Outcome: Number of Tandem Walk Errors at 3 Months and 6 Months
Description: Observed via the Tandem Walk Test at baseline, 3 months, 6 months. Tandem walk errors were the number of errors while walking a four-meter straight line.
  Place a line on the floor marking the distance. The heel of one foot should be touching the tip of the toes of the other foot. Count the number of errors (stepping off the straight line, not putting heel to toe, needing to grab for support, significant body lean). Participants can use an assistive device if they normally use one.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: errors
Arm/Group | Stepping Online | Stepping On 'Usual Care'
Number analyzed (Participants) | 23 | 22
errors
  Baseline (measured pre-randomization) | 4.55 (3.85) | 2.62 (2.80)
  3 Months: number analyzed (Participants) | 23 | 21
  3 Months | 2.10 (3.35) | 6.84 (3.76)
  6 Months: number analyzed (Participants) | 21 | 21
  6 Months | 2.41 (3.11) | 6.48 (4.45)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On 'Usual Care'; at 3 months; Test type: Superiority; p = 0.001, Fisher Exact; Mean Difference (Final Values) = -4.74, 95% CI 2-sided [-6.61 to -2.89]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On 'Usual Care'; at 6 months; Test type: Superiority; p = 0.001, Fisher Exact; Mean Difference (Final Values) = -4.07, 95% CI 2-sided [-6.47 to -1.68]

3. Secondary Outcome: Gait Speed at 3 Months and 6 Months
Description: Observed at baseline, 3 months, 6 months; measured in meters per second over four meters.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Stepping Online | Stepping On 'Usual Care'
Number analyzed (Participants) | 23 | 22
meters per second
  Baseline (measured pre-randomization) | 0.79 (0.25) | 0.83 (0.24)
  3 Months: number analyzed (Participants) | 23 | 21
  3 Months | 0.87 (0.28) | 0.79 (0.21)
  6 Months: number analyzed (Participants) | 21 | 20
  6 Months | 0.89 (0.24) | 0.75 (0.19)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On 'Usual Care'; 3 months; Test type: Superiority; p = 0.05, Fisher Exact; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [0.00 to 0.16]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On 'Usual Care'; 6 months; Test type: Superiority; p = 0.0003, Fisher Exact; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [0.07 to 0.22]

4. Secondary Outcome: Short Physical Performance Battery (SPPB): Total Balance Test
Description: Standing feet together (side by side) for 10 seconds, followed by standing with side of one heel touching the big toe of the other foot (semi-tandem) for 10 seconds, followed by standing with the heel of one foot in front of the toes of the other (tandem) for 10 seconds.
  Participants are scored either 0 or 1 for each balance exercise with a total possible range from 0-3 where higher scores indicate improved balance.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  baseline (measured pre-randomization) | 2.65 (0.65) | 2.32 (0.78)
  3 months: number analyzed (Participants) | 23 | 21
  3 months | 2.60 (0.70) | 2.57 (0.75)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 2.59 (0.73) | 2.64 (0.60)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; 3 months; Test type: Superiority; p = 0.88, Fisher Exact; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.40 to 0.44]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; 6 months; Test type: Superiority; p = 0.83, Fisher Exact; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.48 to 0.37]

5. Secondary Outcome: Short Physical Performance Battery (SPPB): Gait Speed Test
Description: Participant is timed while walking an 8 foot line on the floor.
  Scoring is as follows:
  0 = could not do
  1. = >5.7 sec (<0.43 m/sec)
  2. = 4.1-6.5 sec (0.44-0.60 m/sec)
  3. = 3.2-4.0 (0.61-0.77 m/sec)
  4. = <3.1 sec (>0.78 m/sec)
Time Frame: 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  baseline (measure pre-randomization) | 3.09 (1.04) | 3.18 (0.85)
  3 months: number analyzed (Participants) | 23 | 21
  3 months | 3.25 (1.00) | 3.07 (0.79)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 3.46 (1.02) | 3.12 (0.83)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; 3 months; Test type: Superiority; p = 0.36, Fisher Exact; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.20 to 0.54]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; 6 months; Test type: Superiority; p = 0.14, Fisher Exact; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.11 to 0.77]

6. Secondary Outcome: Short Physical Performance Battery (SPPB): Chair Stand Test
Description: Participant is timed while attempting to stand up and sit down 5 times from a chair without using their arms.
  Scoring is as follows:
  0 = unable
  1. = > 16.7 sec
  2. = 16.6-13.7 sec
  3. = 13.6-11.2 sec
  4. = < 11.1 sec
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  baseline (measure pre-randomization) | 2.26 (1.21) | 2.41 (1.10)
  3 months: number analyzed (Participants) | 23 | 21
  3 months | 2.14 (1.50) | 1.93 (1.18)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 2.51 (1.47) | 2.24 (1.26)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; 3 months; Test type: Superiority; p = 0.52, Fisher Exact; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.43 to 0.85]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; 6 months; Test type: Superiority; p = 0.36, Fisher Exact; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.31 to 0.85]

7. Secondary Outcome: Short Physical Performance Battery (SPPB): Summary Score
Description: The total possible range of scores for the SPPB repeated chair test, gait test, and balance test is 0-12 where higher scores indicate the best performance.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 21
score on a scale
  baseline (measured pre-randomization) | 8.00 (2.30) | 7.91 (1.85)
  3 months | 7.97 (2.59) | 7.58 (2.18)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 8.55 (2.58) | 8.01 (2.05)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; 3 months; Test type: Superiority; p = 0.43, Fisher Exact; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-0.58 to 1.32]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; 6 months; Test type: Superiority; p = 0.26, Fisher Exact; Mean Difference (Final Values) = 0.54, 95% CI 2-sided [-0.42 to 1.49]

8. Secondary Outcome: Falls Behavioral Risk Scale (FaB)
Description: The Falls Behavioral Scale is a list of 24 statements that describe things participants do in everyday life.
  Participants are to circle 'never', 'sometimes', 'often', 'always' or 'doesn't apply'. Scoring is from 1 (never) to 4 (always) and is reported as the average score where higher scores indicate higher mitigation of fall risk.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  baseline (measured pre-randomization) | 2.73 (0.32) | 2.62 (0.28)
  3 month: number analyzed (Participants) | 23 | 21
  3 month | 2.93 (0.74) | 2.68 (0.30)
  6 month: number analyzed (Participants) | 21 | 21
  6 month | 2.72 (0.31) | 2.92 (0.83)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; 3 months; Test type: Superiority; p = 0.16, Fisher Exact; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.09 to 0.61]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; 6 months; Test type: Superiority; p = 0.29, Fisher Exact; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.55 to 0.17]

9. Secondary Outcome: Revised UCLA Loneliness Scale (R-UCLA)
Description: A 3-item scale (adapted, short form of the full 20-item scale) designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. A 3-point Likert scale is used that ask participants to rate each item as either 3 - "I often feel this way", 2 - "I sometimes feel this way", or 1 - "I hardly ever feel this way". Scoring: Items 1-3 are summed and participants are given a composite score of 3-9, with higher scores indicating a greater sense of loneliness.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  baseline (measured pre-randomization) | 4.30 (1.49) | 4.48 (1.66)
  3 Months: number analyzed (Participants) | 23 | 21
  3 Months | 4.28 (1.68) | 4.37 (1.72)
  6 Months: number analyzed (Participants) | 21 | 21
  6 Months | 4.30 (1.92) | 4.11 (1.48)

10. Secondary Outcome: T-Score for Quality of Life Measured by PROMIS Global Mental Health (GMH) Instrument
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) Quality of Life Short Form is a 10-item instrument that measures both Physical (GPH) and Mental (GMH) Health. Each scale is reported as a T-score. The total possible range of scores for GMH is 21.2 - 67.6 where higher scores indicate better quality of life.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  baseline (measured pre-randomization) | 46.89 (5.04) | 47.58 (4.13)
  3 months: number analyzed (Participants) | 23 | 21
  3 months | 47.12 (5.43) | 47.26 (4.55)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 46.61 (5.89) | 46.94 (5.45)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; 3 months; Test type: Superiority; p = 0.91, Fisher Exact; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-2.66 to 2.40]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; 6 months; Test type: Superiority; p = 0.80, Fisher Exact; Mean Difference (Final Values) = -0.33, 95% CI 2-sided [-2.79 to 2.15]

11. Secondary Outcome: T-Score for Quality of Life Measured by PROMIS Global Physical Health (GPH) Instrument
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) Quality of Life Short Form is a 10-item instrument that measures both Physical (GPH) and Mental (GMH) Health. Each scale is reported as a T-score. The total possible range of scores for GPH is 16.2 - 67.7 where higher scores indicate better quality of life.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  baseline (measured pre-randomization) | 42.41 (5.84) | 43.31 (4.66)
  3 months: number analyzed (Participants) | 23 | 21
  3 months | 43.40 (5.60) | 42.77 (4.77)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 43.95 (4.54) | 42.76 (5.74)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; 3 months; Test type: Superiority; p = 0.54, Fisher Exact; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-1.44 to 2.64]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; 6 months; Test type: Superiority; p = 0.38, Fisher Exact; Mean Difference (Final Values) = 1.18, 95% CI 2-sided [-1.49 to 3.81]

12. Secondary Outcome: Physical Activity Barriers Self-Efficacy Score
Description: Self-efficacy to reduce barriers to exercise was measured using a 16-item survey where participants rate their confidence that they could perform falls prevention exercises every day for the next 3 months under various circumstances, from 0% 'not at all confident' to 100% 'very confident'. Scores will be reported from 0-10 with higher scores indicated increased self-efficacy.
Time Frame: up to 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  baseline (measured pre-randomization) | 6.66 (2.53) | 6.43 (1.28)
  3 months | 5.33 (2.08) | 5.38 (2.44)
  6 months | 5.47 (2.37) | 5.57 (2.03)

13. Secondary Outcome: Global Rating of Change Score at 6 Months
Description: Measures self-perceived change in balance, quantifying the extent to which a participant's balance has improved or deteriorated in the over time (past 6 months). A single question asks the participant to rate their change in balance inside their house, and a single question asks patients to rate their change in balance outside of their house. A Likert scare of -7 ("a very great deal worse") to +7 ("a very great deal better") is used to rate this perceived change.
Time Frame: 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  Inside Balance: number analyzed (Participants) | 21 | 21
  Inside Balance | 4.29 (2.63) | 2.40 (3.20)
  Outside Balance: number analyzed (Participants) | 21 | 21
  Outside Balance | 4.05 (2.46) | 2.30 (3.16)
  Strength: number analyzed (Participants) | 21 | 21
  Strength | 3.76 (2.93) | 1.90 (3.32)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; Inside Balance; Test type: Superiority; p = 0.04, Fisher Exact; Mean Difference (Final Values) = 1.89, 95% CI 2-sided [0.06 to 3.71]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; Outside Balance; Test type: Superiority; p = 0.05, Fisher Exact; Mean Difference (Final Values) = 1.75, 95% CI 2-sided [-0.02 to 3.51]
Statistical Analysis 3: Comparison: Stepping Online vs Stepping On Usual Care Control; Strength; Test type: Superiority; p = 0.06, Fisher Exact; Mean Difference (Final Values) = 1.86, 95% CI 2-sided [-0.08 to 3.81]

14. Secondary Outcome: Balance Exercise Adherence at 3 and 6 Months
Description: Adherence was assessed at 3 and 6 months as the number of days balance exercises were performed each week.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
days per week
  Balance Exercises at 3 Months: number analyzed (Participants) | 23 | 21
  Balance Exercises at 3 Months | 4.15 (1.58) | 2.53 (2.08)
  Balance Exercises at 6 Months: number analyzed (Participants) | 21 | 21
  Balance Exercises at 6 Months | 2.91 (2.23) | 1.90 (1.91)
Statistical Analysis 1: Comparison: Stepping Online; Balance Exercises at 3 months; Test type: Superiority; p = 0.003, Fisher Exact; Mean Difference (Final Values) = 1.63, 95% CI 2-sided [0.54 to 2.17]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; Balance Exercises at 6 Months; Test type: Superiority; p = 0.11, Fisher Exact; Mean Difference (Final Values) = 1.01, 95% CI 2-sided [-0.22 to 2.24]

15. Secondary Outcome: Strength Exercise Adherence at 3 and 6 Months
Description: Adherence was assessed at 3 and 6 months as the number of days strength exercises were performed each week.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
days per week
  3 Months: number analyzed (Participants) | 23 | 21
  3 Months | 3.17 (1.43) | 2.11 (1.45)
  6 Months: number analyzed (Participants) | 21 | 20
  6 Months | 2.40 (1.64) | 1.64 (1.40)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; Strength Exercises at 3 months; Test type: Superiority; p = 0.01, Fisher Exact; Mean Difference (Final Values) = 1.06, 95% CI 2-sided [0.23 to 1.89]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; Strength Exercises at 6 months; Test type: Superiority; p = 0.11, Fisher Exact; Mean Difference (Final Values) = 0.75, 95% CI 2-sided [-0.16 to 1.67]

16. Secondary Outcome: Social Bonding Score at 3 Months and 6 Months
Description: Socialization included the 5-item Social Bonding Scale at all timepoints measured as the summed score on a Likert scale of 0 (not at all) to 4 (very much), range 0-20.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  baseline (pre-randomization) | 12.83 (3.51) | 12.57 (4.03)
  3 months: number analyzed (Participants) | 23 | 21
  3 months | 14.07 (4.69) | 13.05 (4.51)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 13.52 (3.97) | 10.92 (4.76)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; 3 months; Test type: Superiority; p = 0.38, Fisher Exact; Mean Difference (Final Values) = 1.02, 95% CI 2-sided [-1.30 to 3.30]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; 6 months; Test type: Superiority; p = 0.02, Fisher Exact; Mean Difference (Final Values) = 2.60, 95% CI 2-sided [0.43 to 4.73]

17. Secondary Outcome: Encouragement to do Exercises Score at 3 Months and 6 Months
Description: Socialization included the feeling Encouraged to Exercise at 3 and 6 months on 1 (very difficult) to 5 (very easy) scale.
Time Frame: up to 6 months
Population: Not all participants completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  3 months: number analyzed (Participants) | 23 | 21
  3 months | 3.61 (1.12) | 3.29 (1.06)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 3.34 (1.16) | 2.72 (0.93)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; 3 months; Test type: Superiority; p = 0.33, Fisher Exact; Mean Difference (Final Values) = 0.32, 95% CI 2-sided [-0.33 to 0.97]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; 6 months; Test type: Superiority; p = 0.06, Fisher Exact; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-0.02 to 1.27]

18. Secondary Outcome: Activities Balance Confidence (ABC) Scale at 3 and 6 Months
Description: The ABC instrument measures the confidence of participants from 0% (no confidence) to 100% (completely confident) for activity in a range of conditions. Scoring is from 0-10 where higher numbers are more confidence.
Time Frame: up to 6 months
Population: Not all participants completed the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stepping Online | Stepping On Usual Care Control
Number analyzed (Participants) | 23 | 22
score on a scale
  baseline (measured pre-randomization) | 7.44 (1.67) | 7.63 (1.42)
  3 months: number analyzed (Participants) | 23 | 21
  3 months | 7.76 (1.59) | 7.13 (1.46)
  6 months: number analyzed (Participants) | 21 | 21
  6 months | 7.65 (1.56) | 7.48 (4.76)
Statistical Analysis 1: Comparison: Stepping Online vs Stepping On Usual Care Control; 3 months; Test type: Superiority; p = 0.06, Fisher Exact; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-0.03 to 1.28]
Statistical Analysis 2: Comparison: Stepping Online vs Stepping On Usual Care Control; Test type: Superiority; p = 0.59, Fisher Exact; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [-0.45 to 0.81]

ADVERSE EVENTS:
Time Frame: up to 6 months
Arm/Group | Stepping Online | Stepping On Usual Care Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 0/23 | 0/22

LIMITATIONS AND CAVEATS:
Limitations include the small sample size. With multiple tests/measures significance might have been by chance. Bonferroni corrections were not performed. Fewer than 30% of the SO graduates who were invited enrolled in the study; these results may not be generalizable to all SO graduates. Lack of access to and comfort with online devices were barriers for some refusers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/89/NCT02774889/Prot_SAP_000.pdf